CLINICAL TRIAL: NCT06641284
Title: Gender-Based Differences in Heart Failure Hospitalizations Among Patients With Heart Failure With Reduced Ejection Fraction Treated With Spironolactone: A Prospective Cohort Study
Brief Title: Gender-Based Differences in Heart Failure Hospitalizations Among Patients With Heart Failure Treated With Spironolactone
Status: Completed | Type: Observational
Sponsor: Ahmad Abdullah Salawi (Other Government)
Responsible Party: Sponsor-Investigator, Ahmad Abdullah Salawi, Associate Professor of Pharmaceutics, University of Jazan
Organization: University of Jazan (Other Government)
Other Study IDs: 2460
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: Heart Failure; Gender; Spironolactone
MeSH Terms: conditions — Heart Failure; Coitus | interventions — Spironolactone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Female Group: Patients identified themselves as females (Apparent gender)
  Interventions: Drug: Spironolactone
- The Male Group: Patients identified themselves as males (Apparent gender)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — All patients will receive Spironolactone as a part of their GDMT for Heart Failure

SUMMARY:
Aldosterone antagonists or mineralocorticoid receptor antagonists (MRAs) are used as therapeutic agents for the management of HF with reduced ejection fraction (HFrEF). Gender-related differences have been described in the regulation of the renin-angiotensin-aldosterone system (RAAS), which is at the core of the pathophysiology of HF. Regarding gender-related differences in the use of MRAs, less is known about the effects of androgens on the RAAS, even though studies have suggested that androgens may increase the RAAS pathway. There are conflicting results because many clinical trials were not specifically designed to investigate gender differences.

DETAILED DESCRIPTION:
The RALES trial investigated the effect of spironolactone on symptomatic HF patients without any difference in treatment benefits between both genders. However, only 30 % of the patients enrolled were females. Another trial investigated the gender-based differences in the treatment of HFpEF patients with spironolactone. The results showed no significant sex differences in clinical endpoints, but a substantial reduction in all-cause mortality was associated with spironolactone use in females but not in males. The utilization of HF pharmacotherapy has been controversial, given recent discoveries presented by the PARAGON-HF trial.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥ 18 years) ambulatory patients of both sexes with a diagnosis of HFrEF (LVEF≤ 40%) and NYHA class II-IV under optimized medical therapy who are presented to the outpatient clinic and started spironolactone at the time of enrollment.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Serum creatinine > 2.5 mg/dL (221 µmol/L) in males and > 2 mg/dL (177 µmol/L) in women (or estimated glomerular filtration rate (eGFR) ≤ 30 mL/minute/1.73 m2)
* Hyperkalemia (serum potassium level > 5 mEq/L)
* Renal transplantation
* Concomitant administration of potent CYP3A inhibitors
* Concomitant administration of potassium supplements or potassium-sparing diuretics
* Disorders of the adrenal glands (such as Addison disease).
* Patients who used MRA in the last 2 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (≥ 18 years) ambulatory patients of both sexes with a diagnosis of HFrEF (LVEF≤ 40%) and NYHA class II-IV under optimized medical therapy who are presented to the outpatient clinic and started spironolactone at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
HF Hospitalization | 6 months after enrollment
  The event of hospitalization due to heart failure.

SECONDARY OUTCOMES:
Hospitalization | 6 months after enrollment
  The event of hospitalization due to any cause.
All-cause mortality | 6 months after enrollment
  The event of mortality due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahd Central Hospital, Al ‘Usaylah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided